CLINICAL TRIAL: NCT06882590
Title: A Brief Compassionate-focused Intervention for Older People with Bipolar Disorder
Brief Title: A Compassionate-focused Intervention for Older People with Bipolar Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Imogen Young, Doctoral Student (Trainee Clinical Psychologist), University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 348011
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder I or II
Keywords: Compassion-Focused Therapy; Older Adults; Rumination; Bipolar Disorder; Guilt; Shame
MeSH Terms: conditions — Rumination Syndrome; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapy participants (Other): Participants to receive the compassionate-focused therapy
  Interventions: Other: Compassionate-focused therapy

INTERVENTIONS:
Other: Compassionate-focused therapy — A 9-session therapy intervention targeting negative thinking, feelings of guilt and shame, and cultivating compassion for self and others.

SUMMARY:
The aim of this study is to determine whether it is feasible to deliver a 9-session compassionate-focused therapy for older people with bipolar disorder. Participants will be asked to complete baseline measures and at post-intervention follow-up (12 weeks and 24 weeks) to understand any potential clinical benefits of the therapy.

DETAILED DESCRIPTION:
The present study will evaluate the feasibility of a compassionate-focused intervention targeting rumination that is specifically tailored for older people with bipolar disorder. In addition to evaluating its feasibility, the study will also investigate whether there are any clinical benefits associated with the intervention, namely, any potential reductions in negative rumination and feelings of guilt and shame. To date, there has been no research evaluating the feasibility of this type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years and above.
* Have a nominated healthcare professional (i.e. GP/Care Coordinator)
* Meet the criteria for a diagnosis of bipolar disorder I or II according to the MINI.
* Score of >57 on Ruminative Response Scale (RRS)
* Be able to provide written informed consent.
* Be able to speak sufficient English to engage in the assessments and intervention.

Exclusion Criteria:

* Currently in an episode of mania or hypomania according to the MINI.
* Experiencing 'severe depression' according to the Hamilton Depression Rating Scale, which equates to a score of over 24.
* MoCA score of <22 to exclude for moderate and severe cognitive impairment.
* Currently receiving psychological therapy.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of therapy sessions attended | The timeframe for number of therapy sessions attended will span the length of intervention; from the first assessment session to final therapy session. The estimated period of time over which the event is assessed is up to 9 weeks.
  The primary outcome of the study is the feasibility of the compassionate-focused intervention, which will be measured using the above metric.
Number of participants who drop-out and at which stage of the intervention | The time frame covers first therapy session to final therapy session. The estimated period of time over which the event is assessed is up to 9 weeks.
  The primary outcome of the study is the feasibility of the compassionate-focused intervention, which will be measured using the above metric.

SECONDARY OUTCOMES:
The Altman Self-Rating Mania Scale | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.
The Bipolar Recovery Questionnaire | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.
The Quality of Life in Bipolar Disorder Questionnaire | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.
Other as Shamer Scale | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.
Guilt and Shame Questionnaire | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.
The Compassionate Engagement and Action Scale | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.
Generalised Anxiety Disorder Questionnaire (GAD-7) | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.
Center for Epidemiologic Studies Depression Scale (CES-D) | Changes in outcome measure scores will be recorded from first baseline, to 12 weeks and 24 weeks follow-up
  Any preliminary potential clinical benefits will be determined using the following outcome measures.

OTHER OUTCOMES:
The MINI International Neuropsychiatric Interview | Eligibility portion of the baseline assessments, prior to the intervention.
  Diagnostic interview for Bipolar I or II.
The Hamilton Depression Rating Scale | Eligibility portion of the baseline assessments, prior to the intervention.
  Assess depression severity.
Ruminative Response Scale | Eligibility portion of the baseline assessments, prior to the intervention.
  Assess levels of rumination.
The Montreal Cognitive Assessment (MOCA) | Eligibility portion of the baseline assessments, prior to the intervention.
  Assessment of cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Manchester Mental Health NHS Foundation Trust, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided